CLINICAL TRIAL: NCT00610337
Title: A Phase IIb, Double-Blind, Randomized, Placebo Controlled, Multicenter Study to Assess the Safety and Efficacy of Intraoperative Epidural Cethrin® in Adult Subjects With Acute Cervical Spinal Cord Injury
Brief Title: Safety and Efficacy of Cethrin® in Adult Subjects With Acute Cervical Spinal Cord Injury
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to a change of sponsor
Sponsor: BioAxone BioSciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALSE-C-01
Record Dates: First submitted 2008-01-15; First posted 2008-02-07 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2010-02

CONDITIONS: Acute Cervical Spinal Cord Injury
MeSH Terms: interventions — exoenzyme C3, Clostridium botulinum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 1 (Placebo Comparator)
  Interventions: Procedure: placebo
- 2 (Experimental): 1mg Cethrin®
  Interventions: Drug: Cethrin® (BA-210)
- 3 (Experimental): 3mg Cethrin®
  Interventions: Drug: Cethrin® (BA-210)
- 4 (Experimental): 6mg Cethrin®
  Interventions: Drug: Cethrin® (BA-210)
- 5 (Experimental): 12mg Cethrin®. Administration of this dose is dependent on data from lower doses.
  Interventions: Drug: Cethrin® (BA-210)
- 6 (Experimental): 18mg Cethrin®. Administration of this dose is dependent on data from lower doses.
  Interventions: Drug: Cethrin® (BA-210)

INTERVENTIONS:
Drug: Cethrin® (BA-210) — Intraoperative epidural administration during spinal decompression surgery
  Other Names: Cethrin®
  Arms: 2; 3; 4; 5; 6
Procedure: placebo — Spinal decompression surgery without administration of Cethrin® BA-210
  Arms: 1

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, Phase IIb study to be conducted in North America and Europe and will include male and female subjects with acute cervical SCI, 18 to 62 years of age, who receive clinical trial material (CTM) within 72 hours of injury.

This study is being undertaken to evaluate and confirm the safety and efficacy of CETHRIN®. This adaptive study has been designed to efficiently identify the safest and most effective dose in Phase IIb which will be evaluated in a future Phase III study. Given the current lack of effective treatments for SCI, an improvement in motor ability or activities of daily living in these subjects would be a great advancement in the treatment of SCI.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the requirements of the study, provide informed consent, agree to the study restrictions, and agree to return for the required assessments
2. Males or females, 18 through 62 years of age, inclusive
3. AIS Grade A, complete injury with the ability to obtain accurate baseline assessment
4. Motor neurological level of C5, C6, or C7
5. Subjects with acute cervical SCI scheduled to receive decompression/stabilization surgery
6. Must be willing and able to participate in study procedures and assessments
7. Must be medically stable
8. If of childbearing potential, women must agree to either of the following for the duration of the 12-month trial: (a) abstinence, or (b) if sexually active, to use one of the following methods of birth control: barrier with spermicide, intrauterine device, birth control hormones, or surgical sterilization
9. Must provide witnessed verbal authorization for use and disclosure of protected health information (PHI)

Exclusion Criteria:

1. Subjects who have participated in a clinical trial involving investigational medications, devices or procedures within 30 days before administration of CTM
2. Subjects who require the use of mechanical ventilation
3. Females with a positive serum pregnancy test
4. Females who are breastfeeding
5. Preexisting SCI
6. Subjects who are unable to receive study medication within 72 hours of injury
7. Subjects with peripheral nerve injury, brachial plexus injury, or multifocal SCI
8. Subjects with injuries that prevent a comprehensive ASIA assessment
9. Complete spinal cord transection
10. Acute SCI because of gun shot or knife wound
11. Subjects who are mentally or medically unstable, or are otherwise unlikely to complete the trial in the judgment of the investigator
12. Subjects who present with history of symptomatic cervical spondylotic myelopathy
13. Subjects with moderate to severe traumatic brain injury with a Glasgow Coma Scale score of less than 14
14. History of multiple sclerosis or other neuromuscular disorder
15. History of an adverse reaction to a fibrin sealant or its human or bovine components
16. Clinically significant neurological, cardiac, respiratory, hepatic, or renal disease
17. History of cancer (except for basal cell carcinoma)
18. Hemophilia or other bleeding abnormality
19. Ankylosing spondylitis
20. Use of insulin therapy to control diabetes mellitus within 6 months of SCI
21. Known immunodeficiency, including human immunodeficiency virus or use of immunosuppressive or cancer chemotherapeutic drugs
22. Body mass index (BMI) of ≥40 kg/m2 at screening (Appendix B includes a table for height and weight to calculate BMI)

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Mean change in ASIA motor score | week 26
Death | 12 months
Serious Adverse Events | 12 months

SECONDARY OUTCOMES:
ASIA Impairment Scale (AIS) grade | Week 4, Week 8, Week 16, Week 26, and Week 52
Total motor score, upper extremity motor score, and lower extremity motor score | Week 4, Week 8, Week 16, Week 26, and Week 52
Neurological motor level (right and left) and motor zone of partial preservation (ZPP) (right and left) | Week 4, Week 8, Week 16, Week 26, and Week 52
Change in motor score within the ZPP (right and left) | Week 4, Week 8, Week 16, Week 26, and Week 52
Spinal cord independence measure (SCIM) total score, subscores and individual items | Week 4, Week 8, Week 16, Week 26, and Week 52
Functional independence measure (FIM) total score, subscores and individual items | Week 4, Week 8, Week 16, Week 26, and Week 52
Adverse events | 12 months